CLINICAL TRIAL: NCT05231083
Title: Transcutaneous Electrical Stimulation of the Genital Nerves (GN) to Improve Erection Dysfunction (ED) in Men: a Pilot Study
Brief Title: Genital Nerves Stimulation for Treatment for Erectile Dysfunction
Acronym: GNS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prof. Dr. med. Marc Possover (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Marc Possover, Director Department of Neuropelveology & Operative Gynecology, Possover International Medical Center AG
Organization: Possover International Medical Center AG (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ED1
Record Dates: First submitted 2021-12-31; First posted 2022-02-09 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Erectile Dysfunction
Keywords: erectile dysfunction; Genital Nerves Stimulation
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Monocebtric randomized unblinded pilote study
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A - 20Hz Stimulation (Experimental): Transcutaneous stimulation of the genital nerves at 20Hz
  Interventions: Device: Genital Nerves Stimulation
- Arm B - 60Hz Stimulation (Experimental): Transcutaneous stimulation of the genital nerves at 60Hz
  Interventions: Device: Genital Nerves Stimulation

INTERVENTIONS:
Device: Genital Nerves Stimulation — Transcutaneous electrical stimulation of the genital nerves using a TENS device and skin adhesive surface electrodes

SUMMARY:
Objectives: To perform pilot study using unilateral transcutaneous electrical stimulation (TENS) on thegenital nerves (dorsal nerve penis and cavernous nerves) for improving of the intracorpereal pressure and full penil erection in men after exclusion neurogenic, endrogenic and earteriogenic disorders. The investigators hypothesize that this therapy will be effective at improving erectile dysfunction (ED).

Material and methods: The study will comprised 20 patients with ED randomized in two groups. Two adhesive skin electrodes are placed, one at the root of the penis and near the pubic symphysis as a cathode, and a second 2-3cm lateral to the penis. Stimulation is delivered for 30 min at the maximal tolerable stimulation amplitude at 210μs pulse width and in one group with a pulse rate at 20Hz, the second group at 60Hz. The penile tumescence and rigidity observed during stimulation are recorded in both groups of patients. Erection Harness Score (EHS) and Quality of Erection Questionnaire (QEQ) are assessed at baseline, immediately after stimulation and 2 weeks after stimulation.

DETAILED DESCRIPTION:
The study is a randomized prospective unblended study. 20 male patients with ED participated to the study. Vulnerable patients, patients with a pacemaker, patients with genital lesions, previous pudendal nerve or genital surgeries, vascular disease or neurological disorders are excluded. Due to the risk of iatrogenic lesions of the erectile nerves, patients suffering from ED secondary to radical prostatectomy are not prime candidates for such a study, however due to the incidence of this etiology and the important impact in the general male population, the investigators decided to include these patients in participants study. The assessment at baseline consistes of a medical history, a neuropelveological workup of the pelvic somatic nerves, pudendal ultrasonography with doppler. Stimulation is performed using a battery powered handled stimulator (N602-1C TENS Elektrostimulator - CH). Monophasic square constant current pulse with a pulse duration of 210 μs. The patients are randomized into two separate groups, a group A with fixed stimulation at 20Hz, a group B with fixed stimulation at 60Hz. Because both genital nerves are located just few millimeters below the skin, stimulation can be achieved using two adhesive skin surface electrodes (diameter 32mm, PALS Platinum, Axelgaard, Lystrup, Denmark), one placed at the root of the penis and in vicinity of the symphysis pubis as a cathode, and a second 2-3cm lateral to the penis. Precautions are taken to ensure good contact between skin and the electrodes, including removal of hairs. Furthermore, the patients are instructed to place the electrodes correctly and to clean the skin before application of the electrodes. The patients are encouraged to set the amplitude as high as tolerable each time when stimulating at home.

Because the different genital nerves may react to different frequency of stimulation , stimulation is delivered for 30 min at the maximal tolerable stimulation amplitude at 210μs pulse width with a pulse rate at 20Hz in patients group A, and at 60Hz in patients group B.

The first transcutaneous stimulation is performed in the presence of MP: The penile tumescence and rigidity observed during stimulation are recorded in both groups of patients. Then stimulation is performed at home at least twice daily for 15 min in each session for a period of 2 weeks. The patients recorde the stimulation amplitude after each session. Erection Harness Score (EHS) and Quality of Erection Questionnaire (QEQ) are assessed for 2 weeks before stimulation, during the 2 weeks of stimulation, and for 2 weeks after the final stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting characteristic symptoms of refractory ED

Exclusion Criteria:

* Patients<18y and >90y

  * Patients who have an implanted pacemaker
  * Vulnerable patients with co-morbid conditions should be excluded from this study. These co-morbid conditions include all pathologies of the cardiovascular system (Angina Pectoris, Infarct, Thrombose, Embolie, Hypertonia), pulmonary system (asthma, COPD, chr. Bronchitis), intestinal system (morbus Crohn, diverticulitis..) and any malignant disease. These co-morbid conditions also include neurologic diseases (i.e., stroke, multiple sclerosis, spinal cord injury), sacral dermal pathological conditions, congenital or other anatomical sacral anomalies (e.g. spina bifida, sacral agenesis, trauma sequelae), mobility deficits, medically complicated/uncontrolled diabetes, fecal motility disorders (fecal incontinence/constipation), chronic pelvic pain, history of recurrent urinary tract infections (UTIs), gross hematuria, prior pelvic/vaginal surgeries (incontinence/prolapse surgeries), pelvic cancer (bladder, colon, cervix, uterus, prostate), deeply infiltrating endometriosis of the pelvic plexus, sacral plexus or of the bladder, Reiter´s syndrome, and pelvic radiation.
  * Patients suffering from other CNS disorders (mental disorders, severe psychological problems, cerebrovascular accident less than 6 months ago).
  * Allergies again skin adhesive electrodes
  * Patients with genital lesions/surgeries, pudendal nerve lesion/surgery or genital surgeries, vascular disease or neurological disorders were excluded. Due to the risk of iatrogenic lesions of the erectile nerves, patients suffering from ED secondary to radical prostatectomy are not prime candidates for such a study, however due to the incidence of this etiology and the important impact in the general male population, we decided to include these patients in our study.

Ages: 19 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 20 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Transcutaneous electrical stimulation of the Genital Nerves for treatment ED | 6 months
  Examining the efficacy of transcutaneous genital nerve stimulation (TENS) in the treatment of ED utilizing the International Index of Erectile Function-15 score:
  A. Erectile function (Q1,2,3,4,5,15): Max score 30 B. Orgasmic function (Q9,19): Max score 10 C: Sexual desire (Q11,12): Max score 10 D: Intercourse satisfaction (Q6,7,8): Max score 15 E: Overall satisfaction (Q13,14): Max Score 10
  IEEFscores <14 out of 39 in domain A (erectile function) may be considered for therapy and referred for specialist investigation.

SECONDARY OUTCOMES:
Quality of erection by using two different frequency of stimulation | 60 months
  The quality of erection by using the Erectile Function-15 score will be compared between two different frequency of stimulation, 20 and 60Hz with following scores:
  A. Erectile function (Q1,2,3,4,5,15): Max score 30 B. Orgasmic function (Q9,19): Max score 10 C: Sexual desire (Q11,12): Max score 10 D: Intercourse satisfaction (Q6,7,8): Max score 15 E: Overall satisfaction (Q13,14): Max Score 10 IEEFscores <14 out of 39 in domain A (erectile function) may be considered for therapy and referred for specialist investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Possover, Principal Investigator — Possover International Medical Center AG
Locations (1):
- Possover, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided